CLINICAL TRIAL: NCT06985537
Title: Efficacy of Ultrasound Guided Intralesional Steroid Injection in Idiopathic Granulomatous Mastitis (IGM)
Brief Title: Steroid Injection in Idiopathic Granulomatous Mastitis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aghapy Ghobrial Reda, Prinicipal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Steroid injection in IGM
Record Dates: First submitted 2024-12-11; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Idiopathic Granulomatous Mastitis
Keywords: Idiopathic GM; intralesional steroid injection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Female diagnosed (clinically and histopatgologically) with IGM not pregnant nor immunocompromised (Other): Ultrasound guided intralesional injection of steroids (Triamicinolone) (40mg/ml ) at site of IGM inflammatory mass after injection of local anesthesia ,once every month and follow up for 6 to 12 months
  Interventions: Drug: Ultrasound guided intralesional Steroids injection (Triamicinolone)

INTERVENTIONS:
Drug: Ultrasound guided intralesional Steroids injection (Triamicinolone) — Radiological guided steroid injection of IGM
  Other Names: Triamicinolone as (epirelefan ) (ciscortine)

SUMMARY:
Granulomatous mastitis (GM) is a non-infectious inflammatory breast condition typically affecting young women, often following breastfeeding. Management of GM often begins with anti-inflammatory medications and antibiotics. Steroids, particularly intralesional corticosteroids, are considered the first-line treatment for GM due to their rapid anti-inflammatory and immunosuppressive effects. Steroids help control symptoms such as painful lumps, swelling, and redness. Steroids' effectiveness in providing symptom relief minimizes the need for more invasive treatments such as surgery.

DETAILED DESCRIPTION:
Granulomatous mastitis (GM) is a rare, non-infectious inflammatory breast condition typically affecting young women within five years of childbirth, often following breastfeeding. Its etiology remains unknown, but histologically, GM is characterized by granulomatous inflammation with the presence of giant cells. Clinically, it presents as a palpable mass, sometimes accompanied by lymph node enlargement, mimicking multifocal breast cancer. The disease may also present with abscesses and fistulas, complicating diagnosis and treatment. Imaging studies such as ultrasound and mammography often reveal irregular masses and hypoechoic nodules, suggesting malignancy. Consequently, biopsy is frequently performed to confirm the diagnosis, revealing chronic lobulitis and granulomas.

Management of GM often begins with anti-inflammatory medications and antibiotics, though these are generally ineffective without proper diagnosis. Steroids, particularly intralesional corticosteroids, are considered the first-line treatment for GM due to their rapid anti-inflammatory and immunosuppressive effects. Steroids help control symptoms such as painful lumps, swelling, and redness. While steroid injections are effective, they can cause side effects like skin atrophy and hypopigmentation, though these are typically temporary and resolve over time. Steroids' effectiveness in providing symptom relief minimizes the need for more invasive treatments such as surgery

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with IGM confirmed clinically and histopathologically , willing to undergo intralesional steroid treatment.

Exclusion Criteria:

* Patients with active infections.
* Patients on immunosuppressive therapy.
* pregnant women.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Clinical Resolution Rate at 12 Weeks Post-Treatment And Reduction in Size | 12 weeks (±1 week) after intralesional steroid injection per participant
  To evaluate the clinical efficacy of intralesional steroid injections in reducing lesion size and resolving symptoms in patients with IGM.
  Anti-inflammatory effect: Steroids like triamcinolone reduce the inflammatory response in breast tissue, alleviating pain, swelling, and mass formation. • Immune modulation: As GM is often immune-mediated, steroids suppress the local immune reaction that drives granuloma formation.
  Anti-inflammatory effect: Steroids like triamcinolone reduce the inflammatory response in the breast tissue, which is the main driver of pain, swelling, and mass formation in GM
  • Immune modulation: Since GM is often immune-mediated, steroids help by suppressing the local immune reaction that is causing granuloma formation.
Clinical Resolution Rate at 12 Weeks Post-Treatment and Reduction in Lesion Size | 12 weeks (±1 week) after intralesional steroid injection per participant
  To evaluate the clinical efficacy of intralesional steroid injections in reducing lesion size and resolving symptoms in patients with IGM.
  Anti-inflammatory effect: Steroids like triamcinolone reduce the inflammatory response in breast tissue, alleviating pain, swelling, and mass formation. • Immune modulation: As GM is often immune-mediated, steroids suppress the local immune reaction that drives granuloma formation.
  help determine whether the therapeutic effect observed at 12 weeks is maintained or further improved by 24 weeks, offering insight into long-term effectiveness and recurrence risk.
  help determine whether the therapeutic effect observed at 12 weeks is maintained or further improved by 24 weeks, offering insight into long-term effectiveness and recurrence risk.
  determine whether the therapeutic effect observed at 12 weeks is maintained or further improved by 24 weeks, offering

REFERENCES:
- [Background] Han BK, Choe YH, Park JM, Moon WK, Ko YH, Yang JH, Nam SJ. Granulomatous mastitis: mammographic and sonographic appearances. AJR Am J Roentgenol. 1999 Aug;173(2):317-20. doi: 10.2214/ajr.173.2.10430126.
- [Background] Toktas O, Konca C, Trabulus DC, Soyder A, Koksal H, Karanlik H, Kamali Polat A, Ozbas S, Yormaz S, Isik A, Sezgin E, Soran A. A Novel First-Line Treatment Alternative for Noncomplicated Idiopathic Granulomatous Mastitis: Combined Intralesional Steroid Injection with Topical Steroid Administration. Breast Care (Basel). 2021 Apr;16(2):181-187. doi: 10.1159/000507951. Epub 2020 Jun 30. PMID 34012373
- [Background] Godazandeh G, Shojaee L, Alizadeh-Navaei R, Hessami A. Corticosteroids in idiopathic granulomatous mastitis: a systematic review and meta-analysis. Surg Today. 2021 Dec;51(12):1897-1905. doi: 10.1007/s00595-021-02234-4. Epub 2021 Feb 15. PMID 33590327
- [Background] Erturk TF, Cakir O, Yaprak Bayrak B, Gunes A, Aydemir S, Utkan NZ. Local Steroid Treatment: An Effective Procedure for Idiopathic Granulomatous Mastitis, Including Complicated Cases. J Invest Surg. 2022 Apr;35(4):745-751. doi: 10.1080/08941939.2021.1933272. Epub 2021 Jun 21. PMID 34154493
- [Background] Tekgoz E, Colak S, Cinar M, Yilmaz S. Treatment of idiopathic granulomatous mastitis and factors related with disease recurrence. Turk J Med Sci. 2020 Aug 26;50(5):1380-1386. doi: 10.3906/sag-2003-93. PMID 32394683
- [Background] Skandarajah A, Marley L. Idiopathic granulomatous mastitis: a medical or surgical disease of the breast? ANZ J Surg. 2015 Dec;85(12):979-82. doi: 10.1111/ans.12929. Epub 2014 Nov 26. PMID 25424519
- [Background] Mizrakli T, Velidedeoglu M, Yemisen M, Mete B, Kilic F, Yilmaz H, Ozturk T, Ozaras R, Aydogan F, Perek A. Corticosteroid treatment in the management of idiopathic granulomatous mastitis to avoid unnecessary surgery. Surg Today. 2015 Apr;45(4):457-65. doi: 10.1007/s00595-014-0966-5. Epub 2014 Jul 4. PMID 24993812
- [Background] Akcan A, Oz AB, Dogan S, Akgun H, Akyuz M, Ok E, Gok M, Talih T. Idiopathic Granulomatous Mastitis: Comparison of Wide Local Excision with or without Corticosteroid Therapy. Breast Care (Basel). 2014 May;9(2):111-5. doi: 10.1159/000360926. PMID 24944554
- [Background] Altintoprak F, Kivilcim T, Yalkin O, Uzunoglu Y, Kahyaoglu Z, Dilek ON. Topical Steroids Are Effective in the Treatment of Idiopathic Granulomatous Mastitis. World J Surg. 2015 Nov;39(11):2718-23. doi: 10.1007/s00268-015-3147-9. PMID 26148520
- [Background] Chirappapha P, Thaweepworadej P, Supsamutchai C, Biadul N, Lertsithichai P. Idiopathic granulomatous mastitis: A retrospective cohort study between 44 patients with different treatment modalities. Ann Med Surg (Lond). 2018 Nov 9;36:162-167. doi: 10.1016/j.amsu.2018.11.001. eCollection 2018 Dec. PMID 30479764